CLINICAL TRIAL: NCT05702931
Title: Safety and Efficacy of Oral Semaglutide in Hyperglycaemic Patients After Renal Transplantation
Brief Title: Semaglutide Treatment for Hyperglycaemia After Renal Transplantation
Acronym: Sema-RTx
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, MD, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-501170-20-00
Record Dates: First submitted 2022-12-23; First posted 2023-01-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hyperglycemia; Renal Transplant Complication Primary Non-Function; Diabetes
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: An investigator-initiated, placebo-controlled, double-blinded, parallel-group, randomised trial.
Who Masked: Participant
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide treated group (Active Comparator): Oral semaglutide once-daily as add-on to standard-of-care for post-transplant hyperglycaemia
  Interventions: Drug: Semaglutide 14 MG [Rybelsus]
- Placebo treated group (Placebo Comparator): Oral placebo once-daily as add-on to standard-of-care for post-transplant hyperglycaemia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide 14 MG [Rybelsus] — At baseline participants will initiate treatment with 3mg of oral semaglutide dosing from weeks 1 to 4. Depending on tolerability the dose will increase to 7 mg daily from weeks 5 to 8 and 14 mg from week 9. Trial medication will be dispensed to subjects for the first time immediately after randomisation and adjusted week 5 and week 9.
  Other Names: Rybelsus
  Arms: Semaglutide treated group
Drug: Placebo — Saline
  Arms: Placebo treated group

SUMMARY:
Background: Post-transplant hyperglycaemia occurs frequently in renal transplant recipients within the first two weeks after transplantation. Standard-of-care is primarily based on insulin treatment with the adherent risk of hypoglycaemia and weight gain. Semaglutide produces an effective lowering of plasma glucose in diabetes patients with chronic kidney disease (CKD) and leads to a reduction in weight and the incidence of hypoglycaemia. The efficacy of semaglutide is untested in renal transplant recipients, and safety concerns remain, primarily on renal graft function.

Objectives: The primary objective is to establish whether tablet semaglutide (Rybelsus) compared with placebo, both as add-on to standard-of-care, is non-inferior in regulating plasma glucose in patients with hyperglycaemia after renal transplantation. Secondary objectives aim to evaluate the effect of tablet semaglutide on renal graft function, weight, use of insulin, cardiovascular parameters and safety parameters (plasma semaglutide concentration, gastrointestinal side effects, dose of immunosuppressants).

Design: An investigator-initiated, placebo-controlled, double-blinded, parallel-group, randomised trial.

Population: Patients (n = 104) with post-transplant hyperglycaemia or type 2 diabetes and an estimated glomerular filtration rate (eGFR) > 15 ml/min/1.73 m2.

Methods: Participants diagnosed with post-transplant hyperglycaemia or type 2 diabetes, 10 to 40 days post-transplant, will be randomised 1:1 to either 14 weeks of tablet semaglutide once daily or placebo both as add-on to standard glucose-lowering therapy. Participants will maintain weekly contact with the clinic during the first five weeks and at two to four weeks intervals during the remaining study period. During the trial, each patient will be monitored according to blood laboratory values with safety assessed at every visit by a nephrologist. Pre-prandial plasma glucose will be measured in the morning and evening to adjust glucose-lowering therapy after consultation with an endocrinologist. Double blinded continuous glucose monitoring (CGM) will be performed for 10-14 days from baseline and at weeks 5, 9, and 13.

Primary endpoint:

- Mean sensor glucose (mmol/L) evaluated by CGM

Key secondary endpoints:

* Incidence of hypoglycaemia
* Body weight (kg)
* Creatinine (μmol/L)
* Daily insulin dose (IE per day)
* Plasma concentration of semaglutide (nmol/L)
* Blood concentrations of cyclosporine and tacrolimus (μg/L)

DETAILED DESCRIPTION:
Introduction:

In renal transplant recipients, hyperglycaemia develops frequently in the immediate period after renal transplantation. Insulin is the primary choice of treatment but carries the adherent risk of hypoglycaemia and weight gain. Tablet semaglutide is a potent glucose-lowering agent that can reduce weight and the incidence of hypoglycaemia. It also has the ability to delay progression of chronic kidney disease (CKD). However, semaglutide is not recommended for renal transplant recipients, as safety and efficacy has yet to be established. The aim of this study is to prove that semaglutide is safe in renal transplant recipients and potentially just as effective as insulin-treatment. We expect that semaglutide can reduce daily insulin-usage and, for a large number of patients, even completely replace insulin as treatment, thereby avoiding the harmful side-effects of this drug.

Objectives:

The primary aim is to establish if tablet semaglutide (Rybelsus) compared with placebo, both as add-on to standard-of-care, is non-inferior in regulating plasma glucose in patients with hyperglycaemia in the immediate weeks after renal transplantation.

Secondary objectives aim to evaluate the effect of tablet semaglutide on renal allograft function, weight, daily use of insulin and safety parameters (plasma semaglutide concentration, gastrointestinal side effects, dose of immunosuppressants).

Background:

Patients developing end-stage renal disease require renal replacement therapy by either haemodialysis, peritoneal dialysis, or renal transplantation. Renal transplantation is considered the best option for renal replacement therapy in terms of both quality of life and cost-effectiveness. However, in the immediate weeks after renal transplantation hyperglycaemia can develop - a condition termed post-transplant hyperglycaemia that is defined by a plasma glucose ≥ 7.0 mmol/L, or 2-h plasma glucose ≥ 11.1 mmol/L after an oral glucose tolerance test. A cohort study of renal transplant recipients (n=319), without pre-transplant diabetes, found that 66% required glucose-lowering treatment when discharge after renal transplantation. The primary reason for hyperglycaemia is high-dose prednisone in combination with surgical stress and other immunosuppressants. The condition post-transplant diabetes mellitus can be diagnosed once the patient is on stable and minimum immune suppressive treatment.

Current guidelines recommend that oral glucose-lowering agents are used for mild hyperglycaemia and insulin for more pronounced hyperglycaemia. Only oral sulfonylureas and dipeptidyl peptidase-4 (DPP-4) inhibitors are permitted for use shortly after renal transplantation. However, sulfonylureas, as with insulin, carry the risk of hypoglycaemia, and DPP-4 inhibitors have only a modest glucose-lowering effect. Therefor insulin treatment is primarily used with the adherent risk of hypoglycaemia, weight gain and the discomfort of daily subcutaneous injections.

Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) are relatively new glucose-lowering agents that effective lowers plasma glucose by enhancing glucose-dependent insulin secretion, regulating postprandial glucagon, and reducing food intake. GLP-1 RAs are not tested prospectively in the renal transplanted population and only two small and retrospective studies have evaluated the safety and efficacy of GLP-1RAs. Here treatment with a GLP-1 RA was associated with a reduced daily insulin dose and lower incidence of hypoglycaemia. Importantly, renal allograft function remained stable with no required adjustment in immunosuppression. In the general diabetes population, the SUSTAIN-6 trial and the PIONEER-6 trial both found that semaglutide yielded a reduction in haemoglobin A1c (HbA1c) and weight. In addition, the SUSTAIN-6 trial found a delay in progression of renal impairment and a lower risk of cardiovascular mortality.

Semaglutide is metabolised by proteolytic cleavage and alterations in renal function are not expected to influence pharmacokinetics. This notion is supported by studies of patients treated with semaglutide where various degrees of renal impairment, including end-stage renal disease, did not influence pharmacokinetics of semaglutide.

Several concerns remain before semaglutide can be used more widely in renal transplanted population. Semaglutide can induce gastrointestinal symptoms (nausea, vomiting, and diarrhoea) that carries a risk of dehydration and gastric paresis that can cause acute kidney injury. Alterations in gastric emptying could change the uptake of immunosuppressive drugs, which in turn can affect renal allograft function.

Study hypothesis:

The investigators expect in the semaglutide group compared to the placebo group to show:

* Similar mean sensor glucose (mmol/L)
* Similar time-in-range (3.9-10.0 mmol/L)
* Reduction in glucose variability
* Reduction in the incidence of hypoglycaemia
* Reduction in daily dose of insulin
* Reduction in weight
* Unaffected renal function of the transplanted kidney
* Unchanged uptake of immunosuppressive medication

Methods and assessments:

Participants diagnosed with post-transplant hyperglycaemia, 10 to 40 days post-transplant, or type 2 diabetes will be randomised 1:1 to either 14 weeks of tablet semaglutide or placebo both as add-on to standard glucose-lowering therapy. Participants will be in weekly contact with the clinic during the first five weeks and with two to four weeks intervals during the remaining study period (Appendix 1). During the trial, each patient will be monitored according to blood laboratory values and with safety assessed at every visit by a nephrologist. Pre-prandial plasma glucose will be measured morning and evening to adjust glucose-lowering therapy in consultation with an endocrinologist. Blinded CGM will be used for 10-14 days from baseline and at weeks 5, 9, and 13.

Questionnaires on gastrointestinal side effects:

Questionnaires on gastrointestinal side effects will be evaluated using the Gastrointestinal symptom rating scale (GSRS). The 15 items in the GSRS questionnaire combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The reliability and validity of the GSRS are well-documented, and norm values for a general population are available.

Continuous glucose monitoring:

A blinded professional Free Style Libre iQ or Dexcom G6/G7 will be used. The sensor is placed on the back of the upper arm and will record interstitial sensor glucose readings every 5-15 min for 10-14 days. The sensor is water-resistant, and no limitations on physical activity exist. CGM data are double blinded. A minium of three CGM-days must be completed for each CGM-period for inclusion in the data analysis.

Blood samples:

Blood samples will be taken at screening (visit 2) and weeks 2, 3, 4, 5, 7, 9, 12, 13, 14 (end of trial). The following laboratory variables will be measured:

* Haemoglobin, leukocytes, platelets
* ALAT, amylase
* Creatinine, urea, sodium, potassium
* C-reactive protein
* Ionised calcium, total phosphate
* Plasma glucose
* Blood cyclosporine (µg/L) and blood tacrolimus (µg/L) At week 1, 5, 9 and 14 following blood samples will be taken
* LDL, HDL, triglycerides, total cholesterol, HbA1c and intact parathyroid hormone

Trial medication:

At baseline participants will initiate treatment with 3mg of oral semaglutide dosing from weeks 1 to 4. Depending on tolerability the dose will increase to 7 mg daily from weeks 5 to 8 and 14 mg from week 9. Trial medication will be dispensed to subjects for the first time immediately after randomisation and adjusted week 5 and week 9.

Glucose-lowering therapy during the study period:

Semaglutide or placebo will be added on top of standard-of-care treatment. Standard-of-care is generally insulin-based treatment, but sulfonylurea may be used. DPP-4 inhibitors are contraindicated during semaglutide treatment. Standard-of-care is not well defined in the renal transplanted population immediately after transplantation. The investigators suggest the following approach:

Study initiation:

Oral semaglutide 3mg or placebo plus standard-of-care defined as:

* If fasting plasma glucose is 7.0-8.4 mmol/L then administration of 0.1 IE/kg (Insulin glargin)
* If fasting plasma glucose is 8.5-9.4 mmol/L then administration of 0.15 IE/kg (Insulin glargin)
* If fasting plasma glucose is 9.5-10.4 mmol/L then administration of 0.25 IE/kg (Insulin glargin)
* If OGTT ≥ 11.0 mmol/L then administration of 0.1 IE/kg (Insulin glargin)

During the study:

Glycaemic monitoring will be performed using pre-prandial plasma glucose (finger prick) in the morning and evening. Based on these measures, and in consultant with an endocrinologist, the glucose-lowering therapy will be adjusted. The glycaemic target is 4-7 mmol/L morning and 6-10 mmol/L evening (both pre-prandial). When increasing semaglutide long-acting insulin is recommended adjusted at the following due to modest effect of semaglutide within the first week. Add-on therapy with sliding scale of fast-acting insulin or sulfonylureas may be added at the discretion of the endocrinologist. At study completion semaglutide and placebo are discontinued and participants returne to standard-of-care.

Reduction in glucose-lowering therapy should be initiated if morning plasma glucose (pre-prandal) < 4 mmol/L 2 out of 3 days or evening plasma glucose (pre-prandial) < 6 mmol/l 2 out of 3 days or if symptomatic hypoglycaemia occurs. Reduction can be performed by the endocrinologist or by the participant. In the study protocol the investigatorsrecommend the following steps but adjustments are at the discretion of the endocrinologist:

Step 1) Patients in Insulin glargine treatment should be reduced by following regime: Firstly reduce by 4 IU of long-acting insulin. If plasma glucose continuously below target reduce by another 4 IU.

Step 2) If plasma glucose is below target and Insulin glargine is < 8 IU, insulin glargine treatment is stopped completely. Secondly, sulfonylurea is stopped.

Step 3) If insulin glargin/sulfonylurea treatment is discontinued and further reductions is required semaglutide is dose reduced from 14mg to 7mg, then from 7mg to 3mg and then from 3mg to 0mg (patient is still required to complete the full study period if glucose-lowering therapy is discontinued).

Statistical evaluation:

The primary endpoint and the secondary endpoints will be reported based on a per protocol analysis with a compliance >80% of the prescribed trial medication. Some secondary endpoints (safety parameters) will be reported based on the intention-to-treat analysis, thus including all randomized participants.

Justification of sample size/power calculation:

The investigators will test the hypothesis if treatment with semaglutide is non-inferior to standard-of-care, with mean sensor glucose (mmol/L) as the primary endpoint in a homogeneous group of renal-transplanted patients with hyperglycaemia. The trial is powered for the primary endpoint, change in mean sensor glucose to assess non-inferiority. The power calculation is based on CGM data from 30 haemodialysis patients with type 2 diabetes that resembles renal transplant recipients with hyperglycaemia as both groups are primarily treated with insulin as standard-of-care. The group of haemodialysis patients are compared with 36 patients with type 2 diabetes and eGFR above 60ml/min/1.73m2 where the majority was treated with without insulin and with antidiabetic medication such as semaglutide.

Sample size calculation is based on a two-sample one-sided t-test with non-inferiority margin of 2mmol/L, expected difference of 0.9 mmol/L, standard deviation of 1.8, power of 90 % and significance level of 5%. This resulted in 47 patients needed in each group, accounting for possible dropout, 10 % expected, a final sample size of 52 patients in each group is needed.

Effect analysis:

Distribution and changes to endpoints will be described and expressed as means± standard error of the mean or median (range or interquartile range) for continues endpoints and frequencies and percentages for categorical endpoints. Comparison of continues outcomes between groups are done by two-sample t-tests if variables are normally distributed, otherwise Wilcoxon sum-rank test is used instead. Comparison of categorical outcomes are done by chi-squared test or fisher's exact test. Repeated measures are compared by mixed regression models. P-values of less than 5 % will be considered statistically significant.

Analysis of safety parameters:

The safety analysis will be performed based on all randomised subjects. A quantitative description of serious and non-serious adverse events will be presented. A qualitative presentation of serious adverse event will be provided.

Feasibility:

Participants will be recruited from Rigshospitalet, Copenhagen; Aarhus, Aarhus University Hospital and Odense, Odense University hospital. Approximately 250 renal transplants are performed in Denmark and we expect with 20-40% will have post-transplant hyperglycaemia 10-15 days after transplantation equivalent to approximately 40 to 80 patients per year. With an aim of 104 included participants the study is expected to last three years.

Ethical considerations:

Semaglutide is well tested in the general diabetes population and not affected by variations in renal function. Participants will be thoroughly monitored throughout the study period to ensure safety. When the trial has ended, concluded and results have been published, participants will be informed of the results of the trial.

The study is registered at ClinicalTrials.gov prior to initiation and the protocol is compliant with the principles of Helsinki Declaration II. The trial will be conducted in compliance with the Good Clinical Practice (GCP) guidelines. A local GCP monitor from the GCP unit at Copenhagen University Hospital, Frederiksberg Hospital will be allocated to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial-related procedures are performed
2. Male or female; age: 18-80 years
3. Diagnosis of post-transplant hyperglycaemia 10 to 40 days after transplantation: Fasting plasma glucose ≥ 7.0 mmol/L or an oral glucose tolerance test with at plasma glucose ≥ 11.1 mmol/L or Pre-transplant type 2 diabetes: Receiving glucose-lowring treatment prior to kidney transplantation
4. An eGFR > 15 ml/min/1.73 m2 10 to 40 days after renal transplantation
5. Subject must be willing and able to comply with trial protocol

Exclusion Criteria:

1. Type 1 diabetes
2. Dialysis
3. High risk immunological transplantation (not including ABO-incompatible or re-transplantation)
4. Early graft rejection (all rejections verified by biopsy, except borderline rejections. Study initiations can begin 5 days after last dose of rejection treatment with methylprednisolone)
5. Chronic pancreatitis/previous acute pancreatitis
6. Known or suspected hypersensitivity to trial or related products
7. Use of DPP-4 inhibitors within five days prior to screening
8. Use of GLP-1RA within 10 days prior to screening
9. Malignancy (except basal cell carcinoma)
10. Inflammatory bowel disease
11. Previous bowel resection
12. Cardiac disease defined as decompensated heart failure (New York Heart Association class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial infarction within the last six months
13. Any acute condition or exacerbation of chronic condition that would in the investigator's opinion interfere with the initial trial visit schedule and procedures.
14. Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant, or are not using adequate contraceptive methods
15. Impaired liver function (plasma ALAT > two times upper reference levels)
16. Elevated amylase (plasma amylase > two times upper reference levels)
17. Untreated proliferative diabetic retinopathy, untreated diabetic macular edema or active conditions of this type that are not under therapeutic control according
18. Any condition that clinically significantly impairs the observation of the fundus or anterior chamber

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean sensor glucose (mmol/L) | 14 weeks
  Mean sensor glucose evaluated by 10 days of CGM obtained at baseline, week 5, week 9 and week 13.

SECONDARY OUTCOMES:
Percentage time in target range (3.9-10.0 mmol/L) | 14 weeks
  Percentage time in target range evaluated by 10-14 days of CGM obtained at baseline, week 5, week 9 and week 13
Percentage time in hypoglycaemia (level 1 [3.0-3.8 mmol/L] and level 2 [below 3.0 mmol/L]) | 14 weeks
  Percentage time in hypoglycaemia evaluated by 10-14 days of CGM obtained at baseline, week 5, week 9 and week 13
Percentage time in hyperglycaemia (level 1 (10.1-13.9 mmol/L) and level 2 (above 13.9 mmol/L) | 14 weeks
  Percentage time in hyperglycaemia evaluated by 10-14 days of CGM obtained at baseline, week 5, week 9 and week 13
Glucose variability (standard deviation [mmol/L] and coefficient of variation [%]) | 14 weeks
  Glucose variability evaluated by 10-14 days of CGM obtained at baseline, week 5, week 9 and week 13
Glucose management indicator (mmol/mol and %) | 14 weeks
  Glucose management indicator evaluated by 10-14 days of CGM obtained at baseline, week 5, week 9 and week 13
HbA1c (mmol/mol) | 14 weeks
  Measured at week 1, 5, 9, and 14
HbA1c (%) | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Body weight (kg) | 14 weeks
  Measure at baseline, week 5, 9 and 14
Body mass index (kg/m2) | 14 weeks
  Measure at baseline, week 5, 9 and 14
Creatinine (μmol/L) | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
eGFR (ml/min/1.73m2) | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Systolic and diastolic blood pressure (mmHg) | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Urinary albumin-to-creatinine ratio (mg/g) | 14 weeks
  Measure at baseline, week 5, 9 and 14
Plasma concentrations of cholesterol | 14 weeks
  Measure at baseline, week 5, 9 and 14
Plasma concentrations of low-density lipoproteins | 14 weeks
  Measure at baseline, week 5, 9 and 14
PPlasma concentrations of high-density lipoproteins | 14 weeks
  Measure at baseline, week 5, 9 and 14
Plasma concentrations of triglycerides | 14 weeks
  Measure at baseline, week 5, 9 and 14
Daily insulin dose (IE per day) | 14 weeks
  Assessed at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Daily dose of immunosuppressant (prednisone, cyclosporine, tacrolimus, mycophenolate mofetile) | 14 weeks
  Assessed at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Plasma concentration of semaglutide (nmol/L) | 14 weeks
  Measure at baseline, week 5, 9 and 14
Dose-corrected plasma concentration of semaglutide (nmol/L) | 14 weeks
  Measure at baseline, week 5, 9 and 14
Plasma insulin (pmol/L) | 14 weeks
  Measure at baseline, week 5, 9 and 14
C-peptide (nmol/L) | 14 weeks
  Measure at baseline, week 5, 9 and 14
Homeostatic model assessment (HOMA) for assessing beta-cell function and insulin 192 resistance | 14 weeks
  Measure at baseline, week 5, 9 and 14
Plasma alanine transaminase (ALAT) (U/L) | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Plasma amylase (U/L) | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Gastrointestinal side effects evaluated using the Gastrointestinal symptom rating scale (GSRS) | 14 weeks
  Assessed at baseline, week 5, 9 and 14. Consist of 15 gastrointestinal symptomes that are each rated on a 7-point scale with 1 being "no discomfort" and 7 being "very severe discomfort".
Incidence of adverse events and serious adverse events | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14
Incidence of self-reported hypoglycaemic episodes | 14 weeks
  Measured at week 2, 3, 4, 5, 7, 9, 12, 13 and 14

CONTACTS AND LOCATIONS:
Locations (1):
- Department og Nephrology and Endocrinology, Rigshospitalet, Copenhagen, Denmark